CLINICAL TRIAL: NCT04095026
Title: A Study of Direct Brain Recording and Stimulation for Memory Enhancement
Brief Title: Study of Direct Brain Recording and Stimulation for Memory Enhancement
Status: Enrolling by invitation | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 150081; 15-N-0081
Record Dates: First submitted 2019-09-14; First posted 2019-09-19 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-06-05

CONDITIONS: Epilepsy
Keywords: Epilepsy; Cognitive Function; Memory; Seizures; Surgery; Natural History
MeSH Terms: conditions — Epilepsy; Seizures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients age >18 years and <= 65 years enrolled in 11-N-0051 Epilepsy Surgery

SUMMARY:
Background:

- Epilepsy is a seizure disorder. Sometimes it is treated with surgery. During surgery, electrodes are placed on or in the brain. Researchers want to learn more about memory and the brain. They want to do tests on people who are having epilepsy surgery.

Objective:

- To learn more about memory and brain function by recording brain cell activity during memory tasks.

Eligibility:

- Adults age 18 - 65 who have medically intractable epilepsy and will have electrodes placed to identify the source of their seizures. They must be currently enrolled in protocol 11-N-0051.

Design:

* Participants may do memory tests before the electrodes are put in, while they are in place, and after surgery. Researchers may stimulate areas of the brain with small pulses of electricity.
* Researchers will start recording brain activity at least 12 hours after electrodes are placed. They will record while participants are awake and asleep. They will record before, during, and after seizures.
* Participants may have up to 3 testing sessions daily over the 1-3 weeks the electrodes are in place. Each session will last 20-60 minutes.
* Participants will play games on a laptop. Sometimes they may use a button or joystick. This can be done in bed in the hospital.
* Participants may be given a list of words and asked to recall them in a short time.
* Participants may be given pairs of items and asked to remember how they are related.
* Participants may be asked to learn their way around a virtual town on the computer. Their eye movements may be tracked by a small camera.

DETAILED DESCRIPTION:
Objective

The primary objectives of this study are (1) to identify biomarkers of successful memory encoding and retrieval, and (2) to identify brain regions that can be stimulated to affect memory performance. The secondary objective is to identify biomarkers that can be used to predict cognitive impairment following resection surgery.

Study Population

One hundred (100) adult subjects with epilepsy who are enrolled in 11-N-0051 Epilepsy Surgery protocol.

Study Design

We plan to enroll individuals with drug resistant epilepsy who are enrolled in a separate protocol, 11-N-0051 Epilepsy Surgery, and who will undergo a neurosurgical procedure in which seizure activity and cognitive functions are mapped using intracranial electrodes in order to guide resection of seizure generating tissue. In this procedure, surgeons place electrodes solely based on clinical consideration with the goal of identifying the seizure focus (or foci) and also for purposes of functional mapping using electrical stimulation.

We propose to administer computerized memory tasks during the intracranial EEG monitoring period. Memory testing may also occur during other patient visits for protocol 11-N-0051. This testing may occur during a pre-surgical outpatient visit or during Phase 1 (pre-implantation) monitoring, to establish baseline memory performance, or after the resection surgery, to identify potential changes in memory performance due to the resection. All testing associated with this protocol will be done during visits or hospitalizations for 11-N-0051, and this protocol involves no additional study visits.

Some memory test sessions will include low-intensity electrical stimulation of the brain using the intracranial electrodes. During these sessions, brain stimulation trials will be interleaved with non- stimulation trials in a randomized fashion.

EEG recordings will be retrospectively analyzed for the presence of biomarkers that correlate with successful memory performance, and test performance will be compared between the stimulation and no-stimulation conditions.

The studies described here are voluntary and for research purpose only. They will not interfere with the clinical evaluation or decision-making process for epilepsy surgery.

Outcome Measures

The primary outcomes are (1) to identify biomarkers of successful memory encoding and retrieval, and (2) to identify brain regions that can be stimulated to affect memory performance. The secondary outcome is to identify biomarkers that can be used to predict cognitive impairment following resection surgery.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible for entry into the study, candidates must meet all the following criteria:

* Be enrolled in 11-N-0051 Epilepsy Surgery.
* Able to give informed consent.
* Age greater than or equal to 18 years and less than or equal to 65 years

EXCLUSION CRITERIA:

Candidates will be excluded if they:

-Have any disability that would limit their ability to perform study tasks that examine memory function.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are considered for this protocol are those with medically intractable epilepsy and currently enrolled in 11-N-0051 Epilepsy Surgery. The patient population for this study is restricted to patients with medically intractable epilepsy because they require surgery for their condition. All participants in this study will require invasive monitoring as part of a clinical evaluation that may lead to subsequent resection of an epileptogenic focus. Enrollment will be equitable among those individuals who meet the inclusion criteria and will not be based on race, ethnicity, or gender.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-10-28 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
to identify biomarkers of successful memory encoding and retrieval | during visits/hospitalizations for 11-N-0051
  We will compare brain recordings during memory encoding for items that are later recalled versus items that are not later recalled. For example, broadband oscillatory activity from electrodes in human temporal lobe has been shown to predict which items are later recalled
to identify brain regions that can be stimulated to enhance memory performance | during visits/hospitalizations for 11-N-0051
  We will correlate task performance across a variety of memory tasks and electrode locations with stimulation parameters (e.g. frequency and amplitude), to identify those brain areas and stimulation parameters that increase task performance.

SECONDARY OUTCOMES:
to identify biomarkers that can be used to predict cognitive impairment following resection surgery | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Kareem A Zaghloul, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
We do plan to share IPD. We will share all IPD that results in a publication on a public repository, as required by most journals. The data will be de-identified and anonymized.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2015-N-0081.html